CLINICAL TRIAL: NCT01533259
Title: A Phase 3B Open-Label Pilot Study to Evaluate Switching From a Regimen Consisting of Raltegravir Plus Emtricitabine/Tenofovir Disoproxil Fumarate Fixed-Dose Combination (FTC/TDF) to the Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Disoproxil Fumarate (EVG/COBI/FTC/TDF) Single-Tablet Regimen (STR) in Virologically Suppressed, HIV-1 Infected Patients
Brief Title: Open-Label Pilot Study to Evaluate Switching From a Regimen Consisting of Raltegravir Plus Emtricitabine/Tenofovir DF Fixed-Dose Combination to the Elvitegravir/Cobicistat/Emtricitabine/Tenofovir DF Single-Tablet Regimen in Virologically Suppressed, HIV-1 Infected Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-236-0123
Record Dates: First submitted 2012-02-02; First posted 2012-02-15 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Acquired Immunodeficiency Syndrome; HIV Infections
Keywords: HIV-1; HIV; Treatment Experienced
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stribild (Experimental): Participants will switch to Stribild for 48 weeks.
  Interventions: Drug: Stribild

INTERVENTIONS:
Drug: Stribild — Elvitegravir (EVG) 150 mg/cobicistat (COBI) 150 mg/emtricitabine (FTC) 200 mg/tenofovir disoproxil fumarate (TDF) 300 mg single-tablet regimen (STR) administered orally once daily with food

SUMMARY:
This study will evaluate the efficacy of Stribild® (elvitegravir/cobicistat/emtricitabine/tenofovir disoproxil fumarate (EVG/COBI/FTC/TDF)) single-tablet regimen (STR) after switching from a regimen consisting of raltegravir plus Truvada® (FTC/TDF) at baseline in maintaining HIV-1 RNA < 50 copies/mL at Week 12 in virologically suppressed, HIV-1 infected adults. This study will also evaluate the safety, tolerability, and efficacy of Stribild over 24 and 48 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and sign a written informed consent form
* Virologically stable on the current first antiretroviral regimen consisting only of raltegravir twice daily plus FTC/TDF continuously for ≥ 6 months preceding the screening visit and

  * have documented undetectable plasma HIV-1 RNA levels ≥ 6 months preceding the screening visit (measured at least twice using the same assay) and
  * have never experienced two consecutive HIV-1 RNA above detectable levels after first achieving a confirmed HIV-1 RNA level below detectable levels on the first regimen
* HIV-1 RNA < 50 copies/mL at the screening visit
* Have a genotype prior to starting initial antiretroviral therapy and have no known resistance to any of the study agents at any time
* Normal ECG
* Hepatic transaminases ≤ 5 x upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 mg/dL
* Adequate hematologic function
* Serum amylase ≤ 5 x ULN
* Estimated glomerular filtration rate ≥ 70 mL/min
* Females of childbearing potential must agree to utilize highly effective contraception methods or be non-heterosexually active, practice sexual abstinence or have a vasectomized partner from screening throughout the duration of the study period and for 30 days following the last dose of study drug
* Females who utilize hormonal contraceptive as one of their birth control methods must have used the same method for at least three months prior to study dosing
* Males must agree to utilize a highly effective method of contraception during heterosexual intercourse from the screening visit, throughout the duration of the study and for 30 days following discontinuation of investigational medicinal product or must be non heterosexually active, practice sexual abstinence, or be vasectomized

Exclusion Criteria:

* New AIDS defining condition diagnosed within the 21 days prior to screening
* Females who are breastfeeding
* Positive serum pregnancy test (female of childbearing potential)
* Individuals with acute or chronic hepatitis B or hepatitis C co-infection
* Individuals experiencing decompensated cirrhosis
* Have an implanted defibrillator or pacemaker
* Current alcohol or substance abuse that would interfere with compliance
* A history of malignancy within the past 5 years or ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous carcinoma
* Active, serious infections requiring parenteral antibiotic or antifungal therapy within 21 days prior to the baseline visit
* Receiving any investigational drugs
* Participation in any other clinical trial without prior approval from the sponsor
* Have been treated with immunosuppressant therapies or chemotherapeutic agents within 3 months of study screening, or expected to receive these agents or systemic steroids during the study
* Any other clinical condition or prior therapy that would make the individual unsuitable for the study or unable to comply with the dosing requirements
* Receiving ongoing therapy or anticipated to need to initiate drugs or herbal/natural supplements during the study that are contraindicated or not recommended for use, including drugs not to be used with Stribild; or individuals with known allergies to the excipients of the Stribild single tablet regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-01; Primary Completion 2012-11 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Huyen Cao, MD, Study Director — Gilead Sciences
Locations (9):
- United States (9):
  - Kaiser Permanente Los Angeles, Los Angeles, California
  - Peter J. Ruane, MD, Inc., Los Angeles, California
  - Anthony Mills MD, Inc, Los Angeles, California
  - Dupont Circle Physician's Group, Washington D.C., District of Columbia
  - Capital Medical Associates, PC, Washington D.C., District of Columbia
  - Orlando Immunology Center, Orlando, Florida
  - Community Research Initiative of New England, Boston, Massachusetts
  - Central Texas Clinical Research, Austin, Texas
  - Gordon E. Crofoot, MD, PA, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at a total of 7 study sites in the United States. The first participant was screened on 31 January 2012. The last study visit occurred on 23 August 2013.
Pre-assignment Details: 58 participants were screened.
Groups:
- Stribild: Switch from existing treatment regimen to Stribild® (elvitegravir (EVG) 150 mg/cobicistat (COBI) 150 mg/emtricitabine (FTC) 200 mg/tenofovir disoproxil fumarate (TDF) 300 mg) single-tablet regiment (STR) once daily for 48 weeks
Period: Overall Study
Arm/Group | Stribild
Started | 48
Completed | 48
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who received at least one dose of study drug.
Groups:
- Stribild: Switch from existing treatment regimen to Stribild (EVG 150 mg/COBI 150 mg/FTC 200 mg/TDF 300 mg) STR once daily for 48 weeks
Arm/Group | Stribild
Number analyzed (Participants) | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 40
  Black or African American | 7
  Asian | 1
Baseline HIV-1 RNA Category [Number; unit: participants]
  < 50 copies/mL | 46
  50 to < 200 copies/mL | 2
CD4 Cell Count [Mean (Standard Deviation); unit: cells/µL] | 711 (265.9)
HIV Disease Status [Number; unit: participants]
  Asymptomatic | 45
  Symptomatic HIV Infection | 1
  AIDS | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 12
Description: The FDA-defined Snapshot algorithm was used, which defines a patient's virologic response status using only the viral load at the predefined time point within an allowed window of time.
Time Frame: Week 12
Population: Full Analysis Set: participants who received at least one dose of study drug and had no major protocol violations of study drug resistance at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stribild
Number analyzed (Participants) | 48
percentage of participants | 100.0 [92.6 to 100.0]

2. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) and Graded Laboratory Abnormalities
Description: This outcome measure assessed the safety and tolerability profile of Stribild. Treatment-emergent adverse events (AEs) and graded laboratory abnormalities occurring from baseline up to 30 days following the last dose of study drug were summarized.
Time Frame: Up to 48 weeks plus 30 days
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Stribild
Number analyzed (Participants) | 48
percentage of participants
  Any AE | 89.6
  Drug-related AE | 25.0
  Grade 3 or higher AE | 4.2
  Serious AE | 2.1
  Any laboratory abnormality | 91.7
  Grade 3 or 4 laboratory abnormality | 4.2

3. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Weeks 24 and 48
Description: as for outcome 1
Time Frame: Weeks 24 and 48
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stribild
Number analyzed (Participants) | 48
percentage of participants
  Week 24 | 100.0 [92.6 to 100.0]
  Week 48 | 100.0 [92.6 to 100.0]

ADVERSE EVENTS:
Time Frame: Up to 48 weeks plus 30 days
Description: Safety Analysis Set
Arm/Group | Stribild
Serious Adverse Events (participants affected / at risk) | 1/48
Other Adverse Events (participants affected / at risk) | 33/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stribild (N=48)
Chest pain (General disorders) | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stribild (N=48)
Diarrhoea (Gastrointestinal disorders) | 5
Fatigue (General disorders) | 5
Seasonal Allergy (Immune system disorders) | 3
Upper respiratory tract infection (Infections and infestations) | 10
Influenza (Infections and infestations) | 4
Folliculitis (Infections and infestations) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3
Bursitis (Musculoskeletal and connective tissue disorders) | 3
Headache (Nervous system disorders) | 4
Hypoaesthesia (Nervous system disorders) | 3
Insomnia (Psychiatric disorders) | 6
Anxiety (Psychiatric disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years